CLINICAL TRIAL: NCT02875041
Title: Non-Invasive TMS Neuromodulation for Enduring Balance & Locomotion Restoration in Parkinson's Disease: A Feasibility and Pilot Study (Locom-TMS)
Brief Title: Non-Invasive TMS Neuromodulation for Enduring Balance & Locomotion Restoration in Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study required back-to-back physical therapy (PT) and TMS Experimental sessions; as our practice move to another building, away from PT
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16-00966
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease
Keywords: rehabilitation; balance
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) MAGSTIM Rapid2 Therapy (Experimental): TMS is a non-invasive device that employs the use of a magnet on the scalp to measure and potentially modulate cortical excitability. The use of TMS for Parkinson's treatment is experimental.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- MAGSTIM Rapid2 Therapy System (Active Comparator): MAGSTIM Rapid2 Therapy System has been FDA cleared for the treatment of refractory depression.
  Interventions: Device: MAGSTIM Rapid2

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS)
  Arms: Transcranial Magnetic Stimulation (TMS) MAGSTIM Rapid2 Therapy
Device: MAGSTIM Rapid2
  Arms: MAGSTIM Rapid2 Therapy System

SUMMARY:
This is a feasibility and exploratory pilot study of adjuvant transcranial magnetic stimulation (TMS) to physical therapy (PT) for locomotion and balance rehabilitation in Parkinson's disease patients.

DETAILED DESCRIPTION:
The primary outcomes will be feasibility of pairing 10 PT training sessions for PB&G with rTMS therapy immediately following PT treatment session. Secondary outcomes will be exploratory, documenting differential clinical effects of two 'active' rTMS compared to 'sham' rTMS, to investigate ability to improve motor and functional recovery outcomes. Outcome measures will be a combination of assessments regularly conducted during PT treatment sessions validated in people with PD (these will doubly serve as our study measures) and several PD oriented outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD confirmed by a neurologist with expertise in movement disorders;
* Hoehn and Yahr stage 2 to 4;
* On L-Dopa and/or Dopamine Agonist daily treatment regimen;
* On a stable medication regimen since at least 2 weeks prior the enrolment in the study and, in the view of the treating neurologist, unlikely to require medication adjustments in the following 3 months;
* Posture, locomotion and balance deficits requiring at least 10 sessions of PT.

Exclusion Criteria:

* History of seizure disorder, including febrile seizures, fainting spells or syncope of unknown cause(s);
* Neurological disorder other than PD including stroke (mild-to-moderate micro vascular disease is allowed), traumatic brain injury, brain tumors, hydrocephalus;
* Major or unstable medical illness;
* Pacemakers, neurostimulators, tattoos or metal foreign bodies in the head area (dental fillings are allowed);
* Untreated depression; or Beck Depression Inventory (BDI)>22
* Taking any of the following medications within the four weeks prior to the start of the study: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, bupropion, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, and theophylline;
* History of moderate or severe dementia, or history of Mini Mental State Examination (MMSE) <20 or Montreal Cognitive Assessment (MoCA) <22;
* Physical therapy treatment contraindications as determined by physiotherapist.

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Mini Balance Evaluation Systems Test | 15 Minutes
  (Mini-BESTest): This is a clinical balance assessment tool that asses dynamic balance through 14 items. It requires 10-15 minutes to be administered. Physical therapists at Rusk use this scale during their normal evaluative sessions.
Five times sit to stand (5XSST) | 5 Minutes
  This is a measure of functional lower limb muscle strength and may be useful in quantifying functional change of transitional movements. Physical therapists use this scale during their normal evaluative sessions. We will use those data collected for our outcome purposes. It requires < 5 minutes to be administered. It is highly recommended and validated in PD by Parkinson's task force PD EDGE.
Timed up and go (TUG): | 3 Minutes
  Assess walking speed in meters per second over a short duration. Time is measured as subject walks a set distance. Physical therapists use this scale during their normal evaluative sessions.
Unified Parkinson's Disease Rating Scale (UPDRS) | 15 Minutes
  The UPDRS is a Parkinson's rating scale which includes evaluations of mentation, behavior, mood, and activities of daily life as well as a clinician scored evaluation to assess motor symptoms of Parkinson's disease.
Clinical Global Impression Scale-Severity and Improvement (CGI-S and CGI-I | 15 Minutes
  CGI was designed to provide a brief stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. Its use has expanded to assess prior to and after any intervention. It takes less than a minute to administer by an experienced rater and it is a great tool to track clinical progress across time.
Parkinson's disease questionnaire-39 (PDQ-39) | 20 Minutes
  Self-report questionnaire that assess PD-specific health related quality over the last month. It assessed how often patients experience difficulties across 8 quality of life dimensions and asses impact of PD on specific dimensions of functioning and well-being. It has become the most frequently used disease-specific measure of health status. It takes 10-20 minutes to be administered.
New Freezing of Gait Questionnaire (NFOG-Q) | 20 Minutes
  This questionnaire will ask questions about symptoms of gait freezing (not being able to move). The NFOG-Q is a reliable tool to detect and evaluate the impact and severity of FOG in PD.

CONTACTS AND LOCATIONS:
Overall Officials: Milton Biagioni, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States